CLINICAL TRIAL: NCT04368962
Title: DSA Risk Factors in Chinese Kidney Transplant Patients Using MPA-based Immunosuppression Protocol: A Multi-center Clinical Study
Brief Title: DSA Risk Factors in MMF-based Immunosuppressed Post-transplanted Patients
Acronym: DRFMBIPTP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2019LSK-038-1
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-08

CONDITIONS: Antibody-mediated Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample to dectect MMF trough concentration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MMF group: Post-transplant patients accept immunosuppression protocol based on MMF for at least 12 months.

SUMMARY:
Kidney transplantation is the best therapy method for patients with uremia. The main factors affecting the long-term survival of the graft were chronic antibody-mediated rejection and the death of the patients. Newborn donor special antibody (DSA) is a major risk factor for chronic antibody-mediated rejection (AMR) and poor transplantation outcomes. Detection of mycophenolate mofetil (MMF) trough concentration can help estimate its exposure. Deficient exposure of MMF can lead to AMR after transplantation surgery. The aim of this study is to estimate the risk factors of one-year DSA after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* years 18-65
* single organ transplantation
* first time to accept kidney transplantation
* Triple immunosuppression protocol based on MMF, tacrolimus and glucocorticoid
* PRA negative before transplantation
* not pregnant for female

Exclusion Criteria:

* Not accept MMF
* multi-organ transplantation
* pregnancy or lactation period female
* mental illness
* past tumor, peptic ulcer, severe cardiopulmonary disease, active liver disease history
* Cannot regular follow up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients after kidney transplantation using triple immunosuppression protocol based on MMF
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
DSA 12 month | 2021.5-2023.5
  newborn DSA in recipient serum in the first 12 month after transplantation

SECONDARY OUTCOMES:
DSA 6 month | 2020.12-2022.12
  newborn DSA in recipient serum in the first 6 month after transplantation
DSA risk factors | 2020.5-2023.5
  risk factors of newborn DSA
MPA-AUC | 2020.5-2023.5
  trough concentration of MMF in recipients' serum
AR | 2020.5-2023.5
  AMR after transplantation
allograft function | 2021.5-2023.5
  serum creatinine and creatinine clearance in 1 year after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang J, Millis JM, Mao Y, Millis MA, Sang X, Zhong S. Voluntary organ donation system adapted to Chinese cultural values and social reality. Liver Transpl. 2015 Apr;21(4):419-22. doi: 10.1002/lt.24069. Epub 2015 Feb 13. PMID 25545626
- [Background] Miettinen J, Perasaari J, Lauronen J, Qvist E, Valta H, Pakarinen M, Merenmies J, Jalanko H. Donor-specific HLA antibodies and graft function in children after renal transplantation. Pediatr Nephrol. 2012 Jun;27(6):1011-9. doi: 10.1007/s00467-012-2101-4. Epub 2011 Oct 13. PMID 21993970
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Ginevri F, Nocera A, Comoli P, Innocente A, Cioni M, Parodi A, Fontana I, Magnasco A, Nocco A, Tagliamacco A, Sementa A, Ceriolo P, Ghio L, Zecca M, Cardillo M, Garibotto G, Ghiggeri GM, Poli F. Posttransplant de novo donor-specific hla antibodies identify pediatric kidney recipients at risk for late antibody-mediated rejection. Am J Transplant. 2012 Dec;12(12):3355-62. doi: 10.1111/j.1600-6143.2012.04251.x. Epub 2012 Sep 7. PMID 22959074
- [Result] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071